CLINICAL TRIAL: NCT07293923
Title: Clinical Feasibility Study of the Magenta Elevate™ Percutaneous Left Ventricular Assist Device (pLVAD) System in Patients With Cardiogenic Shock
Brief Title: Magenta Elevate™ Clinical Feasibility Study in Cardiogenic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magenta Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRD00691
Record Dates: First submitted 2025-11-24; First posted 2025-12-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiogenic Shock; Heart Failure; Acute Myocardial Infarction (AMI)
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiogenic shock (Experimental): Acute myocardial infarction or acutely decompensated heart failure and cardiogenic shock patients
  Interventions: Device: Elevate™ System

INTERVENTIONS:
Device: Elevate™ System — The Elevate™ percutaneous Left Ventricular Assist Device System

SUMMARY:
The Elevate™ CS Clinical Feasibility Study is designed to evaluate the initial safety, effectiveness, and device performance of the Magenta Elevate™ System in patients with cardiogenic shock due to isolated or predominant left ventricular failure.

DETAILED DESCRIPTION:
The Elevate™ CS Clinical Feasibility Study is planned as a prospective, single-arm, interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock of less than 24 hours duration.
* Left ventricular ejection fraction < 45% and > 15%, as determined by echocardiography on the day of inclusion.
* No more than mild right ventricular dysfunction, as determined by echocardiography on the day of inclusion.
* Signed informed consent.

Exclusion Criteria:

* Other causes of shock: hypovolemia, sepsis (any active systemic infection including acute myocarditis), pulmonary embolism or anaphylaxis.
* Patient with oxygen saturation < 90% (pulse oximeter/arterial) at the planned time of device placement (uncorrected by oxygen supplementation or intubation).
* Sustained VT (at the time of the enrollment).
* Significant right heart failure/right ventricular dysfunction.
* Awake patient who is unable to remain in a stable recumbent position due to restlessness or lack of cooperation for other reasons.
* Hypertrophic obstructive cardiomyopathy.
* Left ventricular thrombus.
* Subjects with a placed IABP.
* Mitral and/or aortic valve prothesis, or more than mild native mitral or aortic valve stenosis.
* Aortic valve insufficiency ≥ 2+ (on a 4-grade scale).
* Mechanical complication of myocardial infarction (e.g., ventricular septal rupture, papillary muscle rupture) or evidence of uncorrected Ventricular Septal Defect or Atrial Septal Defect (VSD/ASD).
* Brain damage (e.g., anoxic) or suspected brain damage.
* Stroke or transient ischemic attack within the past 3 months.
* Uncorrectable abnormal coagulation parameters (defined as platelet count < 100,000 or INR > 2.0 or fibrinogen < 1.5 g/L) or active uncontrolled bleeding.
* Allergy, sensitivity or intolerance to heparin, aspirin, Adenosine Diphosphate (ADP) receptor blockers, or contrast media, including known heparin-induced thrombocytopenia.
* Known allergy, sensitivity or intolerance to nickel.
* Known or suspected severe lung disease.
* Evidence of any vascular disease that would preclude placement of the device (e.g., severely calcified and stenosed ilio-femoral vessels).
* Aortic pathology, such as aortic aneurysms, extreme tortuosity, or calcifications that could pose an undue additional risk to the placement of a pLVAD device.
* Any known or suspected disorder causing fragility of blood cells or hemolysis.
* Subject participation in another investigational drug or device trial (post-market registries may be approved by Magenta Medical).
* Life expectancy < 1 year due to comorbidities.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Initial Safety | From device delivery through device removal
  The rate of the composite of Major Device-Related Adverse Events
Device Effectiveness | From baseline to 30 minutes of device activation
  Hemodynamic stability and/or improvement from baseline following device activation, defined as:
  * Number (percentage) of patients with MAP>60mmHg
  * Improvement in MAP
Device Performance | From device delivery through device removal
  * Rate of successful delivery of the Elevate™ System
  * Rate of successful deployment of the Elevate™ System
  * Rate of successful use of the Elevate™ System
  * Rate of successful retrieval of the Elevate™ System

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Lalazar, Study Director — Magenta Medical
Locations (4):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart Center, Tbilisi
- Israel (2):
  - Shamir Medical Center, Be’er Ya‘aqov
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No